CLINICAL TRIAL: NCT00360022
Title: Improving the Transition of Care From Pediatric GI to Adult GI for Patients With IBD: A Prospective Randomized Trial of a New Model
Brief Title: Transition of Inflammatory Bowel Disease (IBD) Patients From Pediatric to Adult Gastroenterologist (GI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problems with subject accrual
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Schwartz, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 060580
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Joint Visits (Experimental): Transition patients will have 2 joint visits performed with the pediatric GI specialist and the adult GI specialist as they transfer care to an adult GI provider.
  Interventions: Other: Joint visits
- Control (No Intervention): Transition patients in the control group will transfer care to adult GI provider in typical manner.

INTERVENTIONS:
Other: Joint visits — Both the pediatric GI specialist and the adult GI specialist will see the patient together at 2 different visits. The first joint visit is lead by the pediatric MD and the second joint visit is lead by the adult MD.
  Arms: Joint Visits

SUMMARY:
The purpose of this study is to determine if the program that has been made to ease the transition of care for adolescent patients with IBD from pediatric gastroenterology to adult gastroenterology is effective to reduce the risk of disease flare during this period. Patient satisfaction with this program will also be assessed.

DETAILED DESCRIPTION:
Approximately 15 to 25% of patients with inflammatory bowel disease are diagnosed prior to the age of 18. The chronic course of this disease means that approximately one quarter of all IBD patients will need to transition from being cared for by a pediatric gastroenterologist to an adult gastroenterologist. Studies in other chronic disease states have identified several problems with the current means of transitioning care from a pediatrician to the adult caregiver including lack of adherence with the proposed treatment, lack of knowledge about the disease, and limited self-care skills. Even without IBD, this can be a time of tremendous turmoil for the adolescent patient. For the chronically ill IBD patient, this stress is further intensified by the underlying illness. Several studies have shown that the risk of flare is increased by non-adherence with medical treatment. The main factors associated with poor adherence include young age and either being under the doctor's care for less than one year or being a new patient for that doctor. Therefore, young adults transferring care from a pediatric gastroenterologist to an adult gastroenterologist are at the highest risk for a bad outcome.

Several recommendations have been published on how to best transition the adolescent IBD patient from pediatric to adult care. The general consensus is that there should be a gradual age specific increase in patient autonomy and involvement in their care prior to being transitioned to an adult gastroenterologist. No study however has incorporated combined clinic visits for the patient with both the pediatric and adult IBD specialist. Furthermore, although these recommendations make logical sense, they have not been assessed objectively.

ELIGIBILITY:
Inclusion Criteria:

A patient may be considered for study participation if all of the following apply:

1. Outpatient of either sex aged ≥ 16 years or older.
2. The patient has a confirmed diagnosis of IBD.
3. No plans to move > 200 miles from Nashville in the subsequent 12 months.
4. The patient has read, understood and signed a written informed consent form. Permission of a minor participant will be obtained via a parent consent form.

Exclusion Criteria:

The patients will be excluded from the study if one or more of the following apply:

1. Unable to give consent.
2. Does not meet inclusion criteria above.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Decrease IBD flare at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David A Schwartz, M.D., Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - The Vanderbilt Clinic, Nashville, Tennessee
  - Vanderbilt Childrens Hospital/ Pediatric Gastroenterology Clinic, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No